CLINICAL TRIAL: NCT03179696
Title: Mobile-Assisted Cognitive Behavior Therapy for Negative Symptoms in Schizophrenia
Acronym: mCBTn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eric Granholm (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Eric Granholm, Professor In Residence, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R61MH110019 (NIH); 1R61MH110019-01 (NIH)
Record Dates: First submitted 2017-05-25; First posted 2017-06-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; CBSST; mobile CBT; negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile-assisted CBT (Experimental): Psychosocial intervention combining in-person and smartphone-based cognitive-behavioral therapy (CBT) for experiential negative symptoms in schizophrenia called, Mobile-assisted Cognitive-Behavioral Therapy for Negative symptoms (mCBTn).
  Interventions: Behavioral: Mobile-assisted CBT

INTERVENTIONS:
Behavioral: Mobile-assisted CBT — mCBTn combines the CBT components that target defeatist attitudes from Cognitive Behavioral Social Skills Training (CBSST) group therapy and mobile smartphone interventions from our prior clinical trials research.

SUMMARY:
This clinical trial will test a combined group therapy plus mobile cognitive behavioral therapy intervention targeting defeatist attitudes in consumers with schizophrenia in order to change motivational negative symptoms linked to defeatist attitudes.

DETAILED DESCRIPTION:
The primary purpose of this project is to test whether a psychosocial intervention, Cognitive Behavioral Social Skills Training (CBSST) combined with a smartphone-based cognitive-behavioral therapy for negative symptoms called, Mobile-assisted Cognitive Behavioral Therapy for Negative Symptoms (mCBTn) can reduce defeatist performance attitudes in consumers with schizophrenia spectrum disorders with persistent moderate-to-severe experiential negative symptoms.The project will also identify the optimal dose to engage the defeatist attitude target. Pupillary responses, an objective psychophysiological biomarker of effort, will be recorded during a cognitive task as a secondary outcome to determine its potential as an end point in clinical trials of motivation and effort.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia or schizoaffective disorder.
* Meets prospective criteria for persistent moderate-to-severe experiential negative symptoms in at least two of the three CAINS Motivation and Pleasure domains (mean of 2 -moderate- or greater for items averaged within the Social, Work or Recreational domains) at the beginning and end of a 2-week evaluation phase.
* Moderate-to-severe defeatist attitudes (DPAS > 50).
* ≥ 6th grade reading level on the Wide Range Achievement Test-4 Reading subtest (needed for reading treatment manual consumer workbook).
* Clinically stable and stable on current medications (no changes within 3 months prior to enrollment and meeting all inclusion/exclusion criteria during longitudinal baseline evaluation at both week -2 and 0).

Exclusion Criteria:

* Prior CBT in the past 2 years.
* Greater than moderate PANSS positive symptoms (P1-Delusions, P2- Disorganization, P3-Hallucinations, or P6-Suspiciousness - any item >5).
* Severe depression on the Calgary Depression Scale for Schizophrenia (CDS >8).
* Extrapyramidal symptoms (Simpson-Angus Scale >7).
* Ocular damage, disease, surgery or medications that affect pupil dilation.
* DSM-5 alcohol or substance use disorder in past 3 months.
* Level of care required interferes with outpatient therapy (e.g., hospitalized; severe medical illness).
* Unable to adequately see or manually manipulate the mobile device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Defeatist performance beliefs (target mechanism) | Assess change from baseline in defeatist performance beliefs at weeks 12, 18 and 24.
  Measure reduction of defeatist performance beliefs severity using the Defeatist Performance Attitude Scale.

SECONDARY OUTCOMES:
Pupillary responses as effort biomarker | Assess change from baseline in pupil dilation at week 12, 18 and 24.
  Measure changes in pupil dilation recorded during a digit span task.
Clinical Assessment Interview for Negative Symptoms (CAINS) | Assess change from baseline in negative symptoms at week 12, 18 and 24.
  Measure changes in motivational negative symptoms on the CAINS.

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Granholm, PhD, Principal Investigator — University of California, San Diego; San Diego Veterans Healthcare System

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buchanan RW. Persistent negative symptoms in schizophrenia: an overview. Schizophr Bull. 2007 Jul;33(4):1013-22. doi: 10.1093/schbul/sbl057. Epub 2006 Nov 10. PMID 17099070
- [Background] Rector NA, Beck AT, Stolar N. The negative symptoms of schizophrenia: a cognitive perspective. Can J Psychiatry. 2005 Apr;50(5):247-57. doi: 10.1177/070674370505000503. PMID 15968839
- [Background] Granholm E, Ben-Zeev D, Link PC, Bradshaw KR, Holden JL. Mobile Assessment and Treatment for Schizophrenia (MATS): a pilot trial of an interactive text-messaging intervention for medication adherence, socialization, and auditory hallucinations. Schizophr Bull. 2012 May;38(3):414-25. doi: 10.1093/schbul/sbr155. Epub 2011 Nov 10. PMID 22080492
- [Background] Granholm E, Holden J, Link PC, McQuaid JR. Randomized clinical trial of cognitive behavioral social skills training for schizophrenia: improvement in functioning and experiential negative symptoms. J Consult Clin Psychol. 2014 Dec;82(6):1173-85. doi: 10.1037/a0037098. Epub 2014 Jun 9. PMID 24911420
- [Background] Granholm E, Ruiz I, Gallegos-Rodriguez Y, Holden J, Link PC. Pupillary Responses as a Biomarker of Diminished Effort Associated With Defeatist Attitudes and Negative Symptoms in Schizophrenia. Biol Psychiatry. 2016 Oct 15;80(8):581-8. doi: 10.1016/j.biopsych.2015.08.037. Epub 2015 Sep 15. PMID 26475673
- [Derived] Granholm E, Holden J, Dwyer K, Mikhael T, Link P, Depp C. Mobile-Assisted Cognitive Behavioral Therapy for Negative Symptoms: Open Single-Arm Trial With Schizophrenia Patients. JMIR Ment Health. 2020 Dec 1;7(12):e24406. doi: 10.2196/24406. PMID 33258792